CLINICAL TRIAL: NCT03144739
Title: Collaborative Child Mental Healthcare in Low-Resource Settings
Brief Title: Collaborative Care for Children's Mental Health Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00111549; R34MH106645-01A1 (NIH)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Depression; Anxiety; Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder; Parent-Child Relations; Substance Use
MeSH Terms: conditions — Depression; Anxiety Disorders; Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: stepped wedge design, hybrid implementation effectiveness
Who Masked: Outcomes Assessor
Masking Description: Research assistants contacting families by telephone for be partially masked - they will not know information about the index child's provider or any baseline characteristics - it will not be possible to completely mask the study phase and thus the control/intervention status of the families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Children enrolled during the control phase will receive care under the Current collaborative care protocol. Participating general practitioners are currently trained to recognize child mental health problems and refer them to partner community mental health centers for treatment.
  Interventions: Other: Current collaborative care protocol
- Intervention (Experimental): Children enrolled during the intervention phase will receive Training in management of children's mental health problems. This will involve treatment by their general practitioner in collaboration with a partner community mental health center; children meeting certain criteria for severity, or whose parents prefer center treatment, will be immediately referred.
  Interventions: Other: Training in management of children's mental health problems

INTERVENTIONS:
Other: Training in management of children's mental health problems — General practitioners will be trained using internationally-developed materials, including the World Health Organization's "mental health need/service gap (mhGAP)" materials and others, adapted for the trial setting (based on formative work that is part of the project). They will be assisted and monitored as part of the ongoing collaborative care program in which they are participating.
  Arms: Intervention
Other: Current collaborative care protocol — General practitioners have been trained to recognize children's mental health problems and to refer them to a partner community mental health center. They receive feedback about the referral but are not encouraged to take on care for the child themselves.
  Arms: Control

SUMMARY:
Background: Mental health problems cause a disproportionate burden of disability among children and youth compared to adults. Primary care plays an important role in efforts to prevent and intervene early in the course of child and adolescent mental health problems. While research with adults has shown the feasibility of integrating mental health care into primary care settings, there have been few studies among children and youth. Evidence remains lacking that integration is feasible in diverse settings, that it improves outcomes, and that methods can be developed to address the mixed symptoms of emerging child/youth problems and their overlap with developmental and parental disorders.

Goals: The purpose of this project is to test the effectiveness of adding a child/youth mental health component into an existing collaborative care program for adult mental health problems. The work will refine a framework for efficient cultural adaption and tailoring of an existing child/youth primary care mental health intervention and then test whether the tailored intervention results in improved child and parent outcomes. The work will also provide evidence about the mechanisms by which those outcomes are achieved and what factors influence uptake of the child/youth component by general practitioners (GPs). These results should be generalizable to low and middle income countries and to underserved areas of the US where there are minimal child mental health resources and family physicians provide the bulk of medical care for children and youth.

Methods: The planned work involves the adaptation/tailoring process followed by a trial with 45 GPs already engaged in collaborative care for adults; the trial will study adding collaborative care for children ages 5-15. GPs will be randomly assigned in groups to begin 6-month control periods involving child mental health screening and referral. They will then receive child/youth training and begin second 6-month periods of screening plus ongoing coaching and booster sessions and collaborative management. Primary outcomes will be measured by recruiting and following for 6 months two cohorts of children/youth and their parents (one control, one collaborative care). Data collected from GPs, parents, youth, and the collaborative care data system will allow measurement of key factors that determine the program's success in helping children and families.

DETAILED DESCRIPTION:
Most mental health problems begin in childhood and adolescence, but delays in receipt of treatment are measured in years to decades. As a result, mental health problems cause a disproportionate burden of disability among children and youth compared to adults, and have a major impact on life course development. Primary care services can play an important role in efforts to prevent and intervene early in the course of child and adolescent mental health problems. Primary care services are widely available and offer an opportunity to interact simultaneously with children and their parents, treat mental health in the context of medical and developmental concerns, and reduce the stigma associated with visiting identifiable mental health facilities. While research with adults has shown the feasibility of integrating mental health care into primary care settings, and that it reduces the burden of mental illnesses, there have been few studies among children and youth and none that address a combined task-shifting/stepped care model. In addition, evidence remains lacking that integration is feasible in diverse settings, that it improves clinical outcomes, and has the potential to be scaled up.

One essential element of integration is "shifting" first-line mental health engagement and treatment tasks to primary care providers. Task shifting requires mental health interventions that fit both the local context of primary care services and the local nature of the problems seen. To date, most adult and child integration models have targeted single conditions at diagnostic levels and relied on additional co-located personnel to provide treatment. To achieve goals of prevention and early intervention, integration models for children and youth must take into account that the symptoms of emerging child and youth problems often suggest multiple possible disorders and can be co-morbid with developmental and parental disorders. By definition, emerging problems amenable to early intervention are likely to be "subthreshold" and not qualify for treatment in a specialty setting, especially when resources are scarce, even though early intervention holds the promise of preventing progression.

The purpose of this trial is to test the effectiveness of adding a child/youth mental health component - tailored to fit the context of primary care into an existing collaborative care program supporting primary care management of adult mental health problems.

The trial's specific aims are to conduct an early-stage hybrid effectiveness-implementation trial with 45 general practitioners in two cities focusing on:

1. Whether delivery of tailored interventions by primary care providers results in improved child and parent mental health outcomes; and exploring the mechanisms by which the interventions achieve those outcomes (which conditions are more likely to be identified and treated, which treatments have the greatest uptake by parents and youth)
2. Whether a coordinated program of training, ongoing coaching, and collaborative care results in uptake of the tailored intervention by primary care providers as evidenced by treatment provided in primary care and participation in collaborative care through consultation and referral.

ELIGIBILITY:
Inclusion Criteria:

* Brought by parent to see general practitioner

Exclusion Criteria:

* Child is acutely physically ill, in acute pain, or general practitioner feels family should not be approached about the study.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Children self-identified or identified by parents as male, female, or other
Enrollment: 1111 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in child mental health-related symptoms | 6 months post enrollment
  Change from baseline to 6-month follow-up on total symptom score of Strengths and Difficulties Questionnaire

SECONDARY OUTCOMES:
Change in child mental health-related functioning | 6 months post enrollment
  Change from baseline to 6-month follow-up on "Impact supplement" score of Strengths and Difficulties Questionnaire
Change in maternal mental health-related symptoms | 6 months post enrollment
  Change from baseline to 6-month follow-up on total score of General Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Wissow, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Will be provided as part of the National Database for Clinical Trials Related to Mental Illness (NDCT)

REFERENCES:
- [Background] Sharifi V, Mojtabai R, Shahrivar Z, Alaghband-Rad J, Zarafshan H, Wissow L. Child and Adolescent Mental Health Care in Iran: Current Status and Future Directions. Arch Iran Med. 2016 Nov;19(11):797-804. PMID 27845550
- [Background] Sharifi V, Shahrivar Z, Zarafshan H, Ashkezary SB, Stuart E, Mojtabai R, Wissow L. Collaborative care for child and youth mental health problems in a middle-income country: study protocol for a randomized controlled trial training general practitioners. Trials. 2019 Jul 8;20(1):405. doi: 10.1186/s13063-019-3467-4. PMID 31287011
- [Derived] Sharifi V, Shahrivar Z, Zarafshan H, Ashezary SB, Arabgol F, Khademi M, Jafarinia M, Hajebi A, Abolhassani F, Emami S, Ashkezari AB, Stuart EA, Mojtabai R, Wissow L. Effect of General Practitioner Training in a Collaborative Child Mental Health Care Program on Children's Mental Health Outcomes in a Low-Resource Setting: A Cluster Randomized Trial. JAMA Psychiatry. 2023 Jan 1;80(1):22-30. doi: 10.1001/jamapsychiatry.2022.3989. PMID 36449318